CLINICAL TRIAL: NCT01216410
Title: The Effect of Adding Metoclopramide and Ondansetron to a Prophylactic Phenylephrine Infusion for the Management of Nausea and Vomiting Associated With Spinal Anesthesia for Cesarean Section
Brief Title: Prevention of Intraoperative Nausea and Vomiting During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00012142; Duke-12142
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2013-03-25 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-07

CONDITIONS: Cesarean Delivery
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Metoclopramide; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Metoclopramide (Active Comparator): Prophylaxis with metoclopramide and phenylephrine infusion.
  Interventions: Drug: Metoclopramide
- Phenylephrine infusion (Placebo Comparator): Prophylactic phenylephrine infusion and placebo antiemetics
  Interventions: Drug: Phenylephrine infusion
- Combination Group (Active Comparator): Metoclopramide and Ondansetron prophylaxis with phenylephrine infusion
  Interventions: Drug: Combination Group

INTERVENTIONS:
Drug: Metoclopramide — Prophylactic Metoclopramide 10 mg given before spinal together with prophylactic phenylephrine infusion
  Arms: Metoclopramide
Drug: Phenylephrine infusion — Prophylactic phenylephrine infusion after spinal and placebo antiemetics
  Arms: Phenylephrine infusion
Drug: Combination Group — Metoclopramide and ondansetron prophylaxis with phenylephrine infusion
  Other Names: Metoclopramide and ondansetron
  Arms: Combination Group

SUMMARY:
The study investigates the incidence of intraoperative nausea and vomiting under spinal anesthesia using a phenylephrine infusion with and without prophylactic antiemetics.

ELIGIBILITY:
Inclusion Criteria:

* English speaking ASA I-II non-laboring women with single gestations ≥36 weeks
* Scheduled or unscheduled cesarean delivery under spinal anesthesia
* Height: 5 feet-5 feet 11 in.

Exclusion Criteria:

* Laboring women needing an emergency cesarean delivery

  * Subjects less than 18 years of age
  * Receipt of a drug with antiemetic properties in the 24 hours prior to cesarean section
  * Allergy to ondansetron, or metoclopramide
  * Severe hypertensive disease of pregnancy defined as systolic blood pressure (SBP)>160mmHg, diastolic blood pressure (DBP)>110mmHg requiring antihypertensive treatment or associated with significant proteinuria.
  * Severe Cardiac disease in pregnancy with marked functional limitations
  * Diabetes type I
  * Patients on Monoamine Oxidase Inhibitors or Tricyclic Antidepressants
  * Morbid obesity (body mass index (BMI)>45)
  * Inclusion in another anesthetic study involving drug administration

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 306 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Habib AS, George RB, McKeen DM, White WD, Ituk US, Megalla SA, Allen TK. Antiemetics added to phenylephrine infusion during cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Mar;121(3):615-623. doi: 10.1097/AOG.0b013e3182839fee. PMID 23635626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 2008-January 2011, University Medical Center
Groups:
- Combination Group: Metoclopramide and Ondansetron prophylaxis
  Combination Group : Metoclopramide and ondansetron prophylaxis
- Metoclopramide: Metoclopramide : Prophylactic Metoclopramide 10 mg given before spinal
- Phenylephrine Infusion: Prophylactic phenylephrine infusion and placebo antiemetics
  Phenylephrine infusion : Prophylactic phenylephrine infusion after spinal
Period: Overall Study
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Started | 103 | 100 | 103
Completed | 101 | 99 | 100
Not Completed | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion | Total
Number analyzed (Participants) | 103 | 100 | 103 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 100 | 103 | 306
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (6) | 31 (5) | 32 (6) | 31 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 100 | 103 | 306
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 55 | 52 | 58 | 165
  Canada | 48 | 48 | 45 | 141

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Nausea and Vomiting
Description: Comparison of intraoperative nausea and vomiting between the 3 groups.
Time Frame: Intraoperatively
Measure: Number; unit: participants
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Number analyzed (Participants) | 101 | 100 | 99
participants | 23 | 31 | 49

2. Secondary Outcome: Postoperative Nausea and Vomiting (PONV)
Time Frame: 0-2h, 2-6h, 6-24h
Measure: Number; unit: participants
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Number analyzed (Participants) | 101 | 99 | 100
participants
  0-2 hrs PONV | 20 | 33 | 39
  2-6 hrs PONV | 28 | 35 | 41
  6-24 hrs PONV | 22 | 26 | 22

3. Secondary Outcome: Pruritus
Time Frame: 0-24 hrs
Measure: Number; unit: participants
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Number analyzed (Participants) | 101 | 99 | 100
participants | 95 | 93 | 97

4. Secondary Outcome: Satisfaction
Description: 1=very satisfied, 2=somewhat satisfied, 3= neither satisfied nor dissatisfied, 4=somewhat dissatisfied, 5= very dissatisfied. Number of very satisfied subjects posted.
Time Frame: 24 h
Measure: Number; unit: participants
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Number analyzed (Participants) | 101 | 99 | 100
participants | 94 | 85 | 87

5. Secondary Outcome: Maternal Hemodynamics
Description: The number of patients with systolic blood pressure decrease to less than 20 % of baseline intraoperatively
Time Frame: Intraoperatively
Measure: Number; unit: participants with SBP< 20 % baseline
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Number analyzed (Participants) | 101 | 99 | 100
participants with SBP< 20 % baseline | 16 | 19 | 16

ADVERSE EVENTS:
Arm/Group | Combination Group | Metoclopramide | Phenylephrine Infusion
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 0/100
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No